CLINICAL TRIAL: NCT01366495
Title: A Randomized Controlled Trial and Cohort Study of HIV Testing and Linkage to Care Corrections
Brief Title: A Randomized Controlled Trial of HIV Testing and Linkage to Care at Community Corrections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R01DA030771-01 (NIH)
Record Dates: First submitted 2011-06-01; First posted 2011-06-06 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: HIV
Keywords: Seek; Test; Treat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- On-site Rapid HIV Testing (Experimental): On-site rapid testing conducted by research staff co-located for the purposes of this study at the probation/parole office.
  Interventions: Behavioral: Project Bridge
- Off-site Referral for HIV Testing (No Intervention): Off-site referral for rapid HIV testing at a community health center or HIV testing clinic
- Project Bridge (Experimental): Project Bridge provides intensive case management for individuals with HIV as they transition back into the community from incarceration. The primary goal of the program is to increase continuity of medical care through social stabilization.
  Interventions: Behavioral: Project Bridge
- Treatment as Usual (No Intervention): Passive referral to HIV community treatment provider.

INTERVENTIONS:
Behavioral: Project Bridge — Project Bridge provides intensive case management for individuals with HIV as they transition back into the community from incarceration. The primary goal of the program is to increase continuity of medical care through social stabilization.
  Arms: On-site Rapid HIV Testing; Project Bridge

SUMMARY:
The investigators propose to conduct both a randomized trial of HIV testing in community corrections, and a randomized trial of linkage to HIV care for people with HIV recruited through community corrections (probation and parole).

DETAILED DESCRIPTION:
The first study is a two-group randomized controlled trial in which 6,000 male and female probationers and parolees in Baltimore City, Maryland and Providence, Rhode Island will be randomly assigned to one of two treatment conditions: 1) On-site rapid testing conducted by research staff co-located for the purposes of this study at the probation/parole office; or 2) Off-site referral for rapid HIV testing at a community health center or HIV testing clinic. Inclusion criteria will be: 1) Adult probationer/parolee; 2) not known to be HIV positive, and 3) resident of greater Baltimore or Providence throughout the study period. Exclusion criteria will be: 1) unable to give informed consent. The second study is a randomized trial, whereby all individuals identified at community corrections with HIV will be offered enrollment in a one-year intervention study to examine the ability to improve linkage into HIV care. Participants will be randomized to receive one of two conditions: 1) Project Bridge for one year, or 2) Treatment as Usual-referral to standard level of care. Moreover, those randomized to TAU will be given an opportunity to "crossover" to PB if they have failed to engage in treatment during the first three months. The rationale for choosing the two cities of Baltimore, MD and Providence, RI is due to the historically high rates of heroin addiction that is associated with multiple HIV-related risk behaviors in these two cities and a high likelihood of being on probation and/or parole. Furthermore, Maryland ranks 10th and Rhode Island ranks 4th in the nation in the number of probationers per 100,000 adult residents.

ELIGIBILITY:
Inclusion Criteria:

1. Probation or Parole;
2. Resident of Baltimore, MD or Providence, RI; 3) Willing to be tested for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2011-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Gordon, D.P.A., Principal Investigator — Friends Research Institute, Inc.; Josiah D Rich, M.D., Principal Investigator — Brown University
Locations (1):
- Maryland Department of Public Safety and Correctional Services (DPSCS), Division of Parole and Probation, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Crable EL, Blue TR, McKenzie M, Rich JD, Gordon MS. Effect of Case Management on HIV Outcomes for Community Corrections Population: Results of an 18-Month Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2021 May 1;87(1):755-762. doi: 10.1097/QAI.0000000000002624. PMID 33492021
- [Derived] Gordon MS, Kinlock TW, McKenzie M, Wilson ME, Rich JD. Rapid HIV testing for individuals on probation/parole: outcomes of an intervention trial. AIDS Behav. 2013 Jul;17(6):2022-30. doi: 10.1007/s10461-013-0456-6. PMID 23536140

RESULTS

PARTICIPANT FLOW:
Groups:
- On-site Testing: HIV testing on-site at probation/parole office
- Off-Site Testing: Off-site HIV testing at a community health center or HIV clinic.
Period: Testing Study
Arm/Group | Project Bridge | Treatment As Usual | On-site Testing | Off-Site Testing
Started | 0 | 0 | 349 | 348
Completed | 0 | 0 | 349 | 348
Not Completed | 0 | 0 | 0 | 0
Period: HIV Study
Arm/Group | Project Bridge | Treatment As Usual | On-site Testing | Off-Site Testing
Started | 50 | 50 | 0 | 0
Completed | 49 | 50 | 0 | 0
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- On-site Testing: Rapid oral swab HIV testing on-site at a community supervision office.
- Off-Site Testing: HIV testing at a community treatment clinic.
- Total: Total of all reporting groups
Arm/Group | Project Bridge | Treatment as Usual | On-site Testing | Off-Site Testing | Total
Number analyzed (Participants) | 50 | 50 | 349 | 348 | 797
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Allows for reporting of two RCT baseline measures.
  years
    HIV Intervention: number analyzed (Participants) | 50 | 50 | 0 | 0 | 100
    HIV Intervention | 46.8 (6.5) | 45.1 (8.6) |  |  | 45.9 (7.6)
    HIV Testing: number analyzed (Participants) | 0 | 0 | 349 | 348 | 697
    HIV Testing |  |  | 39 (11.6) | 38.3 (11.1) | 38.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Allows for reporting of two RCT baseline measures
  Participants
    HIV Intervention: number analyzed (Participants) | 50 | 50 | 0 | 0 | 100
    HIV Intervention: Female | 11 | 11 |  |  | 22
    HIV Intervention: Male | 39 | 39 |  |  | 78
    HIV Testing: number analyzed (Participants) | 0 | 0 | 349 | 348 | 697
    HIV Testing: Female |  |  | 65 | 65 | 130
    HIV Testing: Male |  |  | 284 | 283 | 567
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Allows for reporting of two RCT baseline measures
  Participants
    HIV Intervention: number analyzed (Participants) | 50 | 50 | 0 | 0 | 100
    HIV Intervention: Hispanic or Latino | 1 | 2 |  |  | 3
    HIV Intervention: Not Hispanic or Latino | 49 | 48 |  |  | 97
    HIV Intervention: Unknown or Not Reported | 0 | 0 |  |  | 0
    HIV Testing: number analyzed (Participants) | 0 | 0 | 349 | 348 | 697
    HIV Testing: Hispanic or Latino |  |  | 44 | 51 | 95
    HIV Testing: Not Hispanic or Latino |  |  | 305 | 297 | 602
    HIV Testing: Unknown or Not Reported |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Allows for reporting of two RCT baseline measures
  Participants
    HIV Intervention: number analyzed (Participants) | 50 | 50 | 0 | 0 | 100
    HIV Intervention: American Indian or Alaska Native | 0 | 0 |  |  | 0
    HIV Intervention: Asian | 0 | 0 |  |  | 0
    HIV Intervention: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    HIV Intervention: Black or African American | 47 | 46 |  |  | 93
    HIV Intervention: White | 3 | 4 |  |  | 7
    HIV Intervention: More than one race | 0 | 0 |  |  | 0
    HIV Intervention: Unknown or Not Reported | 0 | 0 |  |  | 0
    HIV Testing: number analyzed (Participants) | 0 | 0 | 349 | 348 | 697
    HIV Testing: American Indian or Alaska Native |  |  | 0 | 0 | 0
    HIV Testing: Asian |  |  | 0 | 0 | 0
    HIV Testing: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    HIV Testing: Black or African American |  |  | 184 | 193 | 377
    HIV Testing: White |  |  | 86 | 89 | 175
    HIV Testing: More than one race |  |  | 0 | 0 | 0
    HIV Testing: Unknown or Not Reported |  |  | 79 | 66 | 145

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Willing to Undergo Rapid HIV Testing
Description: Aim 1: To determine the willingness of the community corrections population to undergo HIV testing (Seek).
  Aim 1a: To compare a strategy of rapid HIV testing on site in community corrections (probation and parole offices) to referral to an off site community HIV testing location with a randomized control study (Test).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | On-site Rapid HIV Testing | Off-site Referral for HIV Testing
Number analyzed (Participants) | 349 | 348
Participants | 318 | 60

2. Primary Outcome: Number of Participants That Entered Community HIV Treatment
Description: Number of Participants That Entered Community HIV Treatment (yes versus no) at the 3-month post baseline follow-up period.
Time Frame: 3-months
Measure: Count of Participants; unit: Participants
Arm/Group | Project Bridge | Treatment As Usual
Number analyzed (Participants) | 49 | 50
Participants | 33 | 35

3. Secondary Outcome: Retention in Community HIV Treatment
Description: Number of Days with Retention in Community HIV Treatment
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Project Bridge | Treatment As Usual
Number analyzed (Participants) | 49 | 50
days | 377.04 (187.44) | 318.82 (208.78)

4. Secondary Outcome: Proportion of Those Prescribed Highly Active Antiretroviral Therapy (HAART) Who Are Undetectable
Description: To determine if a promising, theory driven, case management based strategy (Project Bridge), will be utilized by individuals with HIV recruited through community corrections.
Time Frame: 6,12,18-months
Population: We were unable to obtain official medical records from treatment clinics.
Arm/Group | Project Bridge | Treatment As Usual
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 18-months
Groups:
- Off-site Testing: HIV testing at a community health center or HIV clinic.
Arm/Group | Project Bridge | Treatment As Usual | On-site Testing | Off-site Testing
All-Cause Mortality (participants affected / at risk) | 1/50 | 0/50 | 0/349 | 0/348
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/50 | 0/349 | 0/348
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/349 | 0/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Project Bridge (N=50) | Treatment As Usual (N=50) | On-site Testing (N=349) | Off-site Testing (N=348)
Death (Social circumstances) | 1 (1) | 0 (0) | NA | NA — overdose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes